CLINICAL TRIAL: NCT04969731
Title: An Open-label, Randomized, Multi-center, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Adjuvant Immuncell-LC Therapy Combined With Gemcitabine Versus Adjuvant Gemcitabine Single Therapy After Resection in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: Safety and Efficacy of Immuncell-LC With Gemcitabine in Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILC-P3-PAN
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Adjuvant Therapy; Immuncell-LC; Gemcitabine; ILC-P3-PAN; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immuncell-LC/Gemcitabine (Experimental): Patients will receive 6 cycles Gemcitabine (1000 mg/m2 on Days 1, 8, 15, 28-day a cycle) and Immuncell-LC 16 times during 60 weeks (4 treatments once a week, followed by 4 treatments every other week, then 4 treatments every 4 weeks, and finally 4 treatments every 8 weeks)
  Interventions: Drug: Immuncell-LC; Drug: Gemcitabine
- Gemcitabine (Active Comparator): Patients will receive 6 cycles Gemcitabine alone (1000 mg/m2 on Days 1, 8, 15, 28-day a cycle)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Immuncell-LC — IV
  Other Names: Autologous activated T lymphocyte
  Arms: Immuncell-LC/Gemcitabine
Drug: Gemcitabine — IV

SUMMARY:
PURPOSE: This phase III clinical trial evaluates the efficacy and safety of adjuvant Immuncell-LC therapy combined with gemcitabine versus adjuvant gemcitabine single therapy after R0 or R1 resection in patients with pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
Open-label, Randomized, Multi-center, Parallel, Phase III Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=20 years old, </=80 years old.
2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma that fulfill the following requirements:

   * Participants have undergone a radical full resection (R0) or boundary resection (R1) operation and has elapsed at least two weeks after the resection based on the baseline, up to 12 weeks.
   * Noncancerous ascites.
   * No evidence of distant metastasis (such as liver, peritoneum)
   * No evidence of distant metastasis in other distant abdominal or extra-abdominal organs
   * Scheduled to be given gemcitabine alone as postoperative adjuvant chemotherapy
3. Eastern Cooperative Oncology Group-performance status (ECOG-PS) 0 - 2
4. Life expectancy is at least 12 weeks.
5. Adequate organ and marrow function at the screening and baseline as defined below:

   * Absolute neutrophil count ≥ 1,500/μL
   * Hemoglobin level ≥ 9 g/dL
   * Platelet count ≥ 100,000/μL
   * BUN, serum creatinine ≤ 1.5 × institutional upper limit of normal (ULN)
   * AST, ALT ≤ 2.5 × institutional upper limit of normal (ULN)
   * PT (INR), activated partial thromboplastin time (aPTT) ≤ 1.5 × institutional upper limit of normal (ULN)
6. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Received anticancer therapy including chemotherapy, biological therapy, immunotherapy, hormone therapy, radiation therapy, and other anti-cancer treatments. Note: Neo-adjuvant therapy for pancreatic cancer is allowed.
2. Measurable lesions identified in the pancreas after surgery.
3. Known history at the screening as defined below.

   * Confirmed cases of acquired immunodeficiency, which can be exacerbated by immunotherapy.
   * History of autoimmune diseases that can be exacerbated by immunotherapy. (e.g. rheumatoid arthritis, systemic lupus, vascular inflammation, multiple sclerosis, adolescent-induced insulin-dependent diabetes, T-cell lymphoma, etc.)
   * Active hepatitis B or hepatitis C virus infection confirmed.
   * Human immunodeficiency virus (HIV) antibody test results are positive during screening
   * History of malignant tumors other than pancreatic cancer within five years of screening. Note: skin basal cell cancer/squamous cell cancer, local prostate cancer, thyroid papillary cancer or cervical epithelial cancer can be participated even if 5 years have passed since successful treatment.
4. Known associated disease at the screening as defined below.

   * Severe nephropathy: estimated glomerular filtration rate (eGFR)‡ <30 mL/min/1.73 m2
   * Chest X-ray shows epileptic pneumonia or pulmonary fibrosis with clear, clinical symptoms.
   * Severe infections or other uncontrolled active infectious diseases requiring the administration of antibiotics, antibacterial drugs, antifungal drugs, antiviral drugs, etc. that may affect safety and validity evaluation during clinical trials, as determined by the tester.
   * Holder of thromboembolic disease or bleeding diatheses
   * Those who are deemed unfit to participate in clinical trials because they are not controlled or require treatment (e.g., heart disease, pulmonary dysfunction, renal dysfunction, low blood pressure, hypertension, bone marrow inhibition, liver metastasis, hepatitis, history of alcoholism, myocardial infarction, etc.)
5. Received Immuncell-LC, Natural Killer (NK) cell therapy or other cell therapy drugs within three years prior to screening.
6. Anaphylaxis to the main ingredient or sub-brothers of Immuncell-LC or Gemcitabine
7. Patients who cannot collect blood for manufacturing Immuncell-LC depending on the investigator's judgment.
8. Pregnant or lactating women
9. Fertility women and men who are not willing to use appropriate contraception from screening to 24 weeks after final administration of Immuncell-LC and/or Gemgitabine
10. Received or applied with another investigational products or investigational device within 4 weeks prior to signing a written informed consent document.
11. Patients who are inappropriate or impossible to participate in the trial due to non-recovery of resection or prior chemotherapy depending on the investigator's judgment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) by independent review | Up to approximately 36 months after Last Patient In
  Recurrence free survival is defined as the time from randomization to the date of the recurrence confirmed by independent reviewer

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 36 months after Last Patient In
  Overall survival is defined as the time from randomization to death due to any cause.
Recurrence free survival (RFS) by investigator | Up to approximately 36 months after Last Patient In
  Recurrence free survival is defined as the time from randomization to the date of the recurrence confirmed by investigator
Carbohydrate antigen 19-9 level | Up to approximately 36 months after Last Patient In
  Carbohydrate antigen 19-9 level
Quality of Life (QoL) EORTC QLQ-C30 | Up to approximately 36 months after Last Patient In
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Quality of Life (QoL) EORTC QLQ-PAN26 | Up to approximately 36 months after Last Patient In
  The module comprises 26 questions assessing pain, dietary changes, jaundice, altered bowel habit, emotional problems related to pancreatic cancer, and other symptoms (cachexia, indigestion, flatulence, dry mouth, taste changes). The answers range is the following: not at all - 1 point, a little - 2 points, quite a bit - 3 points, very much - 4 points. Minimum score is 26, maximum is 106. The higher total score represents the worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehak-ro, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi JH, Nam GH, Hong JM, Cho IR, Paik WH, Ryu JK, Kim YT, Lee SH. Cytokine-Induced Killer Cell Immunotherapy Combined With Gemcitabine Reduces Systemic Metastasis in Pancreatic Cancer: An Analysis Using Preclinical Adjuvant Therapy-Mimicking Pancreatic Cancer Xenograft Model. Pancreas. 2022 Oct 1;51(9):1251-1257. doi: 10.1097/MPA.0000000000002176. PMID 37078953